CLINICAL TRIAL: NCT05271591
Title: Generalizability of the REDUCE-IT Results to People of South Asian Descent With Known Atherosclerotic Cardiovascular Disease Living in Canada
Brief Title: Generalizability of REDUCE-IT Results to People of South Asian Descent With Atherosclerotic Cardiovascular Disease in Canada (REDUCE-IT Canada SA)
Status: Completed | Type: Observational
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: HLS Therapeutics, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00061124
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Atherosclerotic Cardiovascular Disease; Myocardial Infarction; Coronary Heart Disease
Keywords: Icosapent Ethyl; Ethnic Origin
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Myocardial Infarction; Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The REDUCE-IT Canada SA Study is a cross-sectional study aiming to determine the proportion of study participants who meet the Health Canada-approved indication for icosapent ethyl (IPE;Vascepa®).

DETAILED DESCRIPTION:
Global derived data indicate that compared to most ethnicities, people of South Asian (SA) descent shoulder a heavier burden and mortality rate for atherosclerotic cardiovascular disease (ASCVD). They are younger at the time of first hospitalization for heart failure and exhibit more high-risk features upon discharge. Canadian data indicate that SAs presented to the hospital later during acute myocardial infarction and are more likely to have an anterior location of infarction. They also tend to be younger at the time of cardiac catheterization than those of European descent and are more likely to have significant left main, multivessel, and distal coronary artery disease. SAs appear to have comparatively pro-atherosclerotic lipid profiles - more small dense LDL particles, lower HDL-C levels, and hypertriglyceridemia - and demonstrate a higher prevalence of diabetes, metabolic syndrome, central adiposity and inflammation.

People of SA descent are markedly underrepresented in clinical trials, and it remains unclear as to whether many of the life-saving therapies are generalizable to this population. The REDUCE-IT Canada SA Study aims to determine the generalizability of the REDUCE-IT study results to people of South Asian descent with known ASCVD living in Canada. Specifically, the study will ascertain the proportion of South Asian individuals that meet the Health Canada indication for IPE; the alignment of the participants' baseline characteristics with those of the REDUCE-IT cohort; the proportion of study participants who have access to private and/or public coverage.

ELIGIBILITY:
Inclusion Criteria:

* Adults 45 years of age or older of SA descent i. A person of SA descent is any individual who self-identifies as Anglo-Indian, Bangladeshi, Bengali, Bhutanese, Goan, Gujarati, Indian, Jatt, Kashmiri, Maharashtrian, Malayali, Nepali, Pakistani, Punjabi, Sindhi, Sinhalese, Sri Lankan, Tamil, Telugu, or other SA descent
* History of ASCVD within the preceding 10 years defined as:

  i. Documented CAD (defined as having experienced a prior MI, coronary artery bypass grafting, percutaneous coronary intervention) ii. Documented cerebrovascular disease (defined as having experienced a prior stroke, transient ischemic attack or carotid revascularization) iii. Documented peripheral artery disease (ankle-brachial index <0.9, or peripheral revascularization)
* On stable statin therapy
* Has had routine bloodwork within 3 years prior to enrolment- Willing and able to provide verbal or written informed consent

Exclusion Criteria:

* Severe congestive heart failure (as defined by New York Heart Association Class IV)
* Any life-threatening disease expected to result in death within the next 2 years
* Any malignancy not considered cured (except basal cell carcinoma of the skin) An individual is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening
* Known severe liver disease
* Known acquired immunodeficiency syndrome such as human immunodeficiency virus infection
* Use of omega-3 fatty acid supplements, fish oil, or icosapent ethyl

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from primary care and cardiology outpatient clinics in the Greater Toronto Area using paper-based and electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Proportion of study participants who meet the Health Canada-approved indication for icosapent ethyl [Product Monograph dated Dec 30, 2019] | 8 weeks

SECONDARY OUTCOMES:
Proportion of study participants whose demographic and biochemical data align with the corresponding baseline criteria of the REDUCE-IT cohort | 8 weeks
Proportion of study participants who have access to private and/or public coverage | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (5):
- Canada (5):
  - Scarborough Health Network, Ajax, Ontario
  - Fenton Medical Centre, Markham, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Legacy Medical Centre, Scarborough Village, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta M. Addressing atherosclerotic cardiovascular disease risk in South Asians: A daunting task ahead. Atherosclerosis. 2020 Dec;315:76-78. doi: 10.1016/j.atherosclerosis.2020.10.892. Epub 2020 Nov 4. No abstract available. PMID 33172687
- [Background] Statistics Canada. Canada [Country] and Ontario [Province] (table). Census Profile. 2016 Census.2017 January 29, 2022. Available from: https://www12.statcan.gc.ca/census-recensement/2016/dp-pd/prof/index.cfm?Lang=E.
- [Background] Enas EA, Garg A, Davidson MA, Nair VM, Huet BA, Yusuf S. Coronary heart disease and its risk factors in first-generation immigrant Asian Indians to the United States of America. Indian Heart J. 1996 Jul-Aug;48(4):343-53. PMID 8908818
- [Background] McKeigue PM, Marmot MG. Mortality from coronary heart disease in Asian communities in London. BMJ. 1988 Oct 8;297(6653):903. doi: 10.1136/bmj.297.6653.903. No abstract available. PMID 3140974
- [Background] Balarajan R. Ethnic differences in mortality from ischaemic heart disease and cerebrovascular disease in England and Wales. BMJ. 1991 Mar 9;302(6776):560-4. doi: 10.1136/bmj.302.6776.560. PMID 2021718
- [Background] Enas EA, Yusuf S, Mehta JL. Prevalence of coronary artery disease in Asian Indians. Am J Cardiol. 1992 Oct 1;70(9):945-9. doi: 10.1016/0002-9149(92)90744-j. No abstract available. PMID 1529952
- [Background] Superko HR, Enas EA, Kotha P, Bhat NK, Garrett B. High-density lipoprotein subclass distribution in individuals of Asian Indian descent: the National Asian Indian Heart Disease Project. Prev Cardiol. 2005 Spring;8(2):81-6. doi: 10.1111/j.1520-037x.2005.3766.x. PMID 15860982
- [Background] Bhardwaj S, Misra A, Misra R, Goel K, Bhatt SP, Rastogi K, Vikram NK, Gulati S. High prevalence of abdominal, intra-abdominal and subcutaneous adiposity and clustering of risk factors among urban Asian Indians in North India. PLoS One. 2011;6(9):e24362. doi: 10.1371/journal.pone.0024362. Epub 2011 Sep 20. PMID 21949711
- [Background] Banerjee AT, Shah B. One Size Does Not Fit All: Diabetes Prevalence Among Immigrants of the South Asian Diaspora. J Immigr Minor Health. 2021 Aug;23(4):653-658. doi: 10.1007/s10903-020-01093-4. Epub 2020 Sep 29. PMID 32990901
- [Derived] Krishnaraj A, Bakbak E, Teoh H, Bhatt DL, Quan A, Puar P, Lambotharan B, Kirubaharan A, Firoz IN, Meglis G, Yanagawa B, Bari B, Kirubaharan R, Vijayaraghavan R, Hess DA, Demchuk AM, Mancini GBJ, Tanguay JF, Tardif JC, Voisine P, Leiter LA, Verma S. Generalizability of the REDUCE-IT trial to South Asians with cardiovascular disease. Med. 2023 Feb 10;4(2):130-138.e1. doi: 10.1016/j.medj.2022.12.008. Epub 2023 Jan 10. PMID 36630964